CLINICAL TRIAL: NCT04712422
Title: Poor Neck Proprioception May Cause Balance Deficits in Myotonic Dystrophy 1
Acronym: CABLAMYD
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Fondazione Serena Onlus - Centro Clinico NeMO Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 24C020
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Myotonic Dystrophy 1
Keywords: Myotonic Dystrophy 1; Accidental falls; Ataxia; Postural balance; Rehabilitation
MeSH Terms: conditions — Myotonic Dystrophy; Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: At least 25 healthy participants aged from 18 to 50 years old. Participants will be excluded if pregnant.
  Interventions: Other: Healthy subjects
- Pathologic group: At least 22 participants with diagnosis of Myotonic Dystrophy 1.
  Interventions: Other: Pathologic group

INTERVENTIONS:
Other: Healthy subjects — Participants will be tested for their foot dominance by means of the Waterloo footedness questionnaire-revised, their hand dominance by means of the Edinburgh inventory, and their eyedness Coren's Lateral Preference Inventory.
  Participants will perform a cervical repositioning test. They will seat in a chair in front of a Plexiglas screen with the eye closed. The operator will guide the participant in four positions: at 30° right/left rotation and at 25° extension/flexion. The participant will be then asked to reproduce the angle. Each movement will be repeated four times in a random order. The whole sequence will be repeated by another second operator. Both the tests will be repeated after two weeks.
  Head movements will be detected using an optoelectronic system using passive markers positioned on the head of the participant.
  Groups: Healthy participants
Other: Pathologic group — Clinical evaluation of the participants will be performed by means of the Myotonic Dystrophy Health Index (MDHI), the Rivermead Mobility Index (RMI), the Fall Events Questionnaire, and the Dizziness Handicap Inventory- short form (DHIsf).
  Participants will perform a cervical repositioning test. Participants will seat in a chair in front of a Plexiglas screen with the eye closed. The operator will guide the participant in four positions: at 30° right/left rotation and at 25° extension/flexion. The participant will be then asked to reproduce the angle. Each movement will be repeated four times in a random order.
  Head movements will be detected using an optoelectronic system using passive markers positioned on the head of the participant.
  Participants will then perform test of balance in standing, using the EquiTest platform. Individuals will be requested to perform three different tasks: sensory organization test, adaptation test-upward tilt, and adaptation test-downward tilt.
  Groups: Pathologic group

SUMMARY:
Impairment of balance and gait are frequent complaints in patients with myotonic dystrophy type 1 (DM1). In these persons, there is an increased risk for stumbles and falls when compared to normal subjects. An underestimated cause of falls might be the weakness of neck flexor muscles (due to cervical ataxia). It is well known that fibres of muscle spindles are receptors combining a specialized sub-set of muscle fibers with a specialized array of both sensory and motor nerve fibers. Spindles transduce into neural afferent discharges the muscle length and length changes. They are very dense in deep neck muscles, are crucial to body balance and gage orientation, and are severely affected in DM1. Preliminary results suggest that falls could reflect imbalance. These indicate that cervical ataxia may come into play because of muscle spindle fibre disruption. In light of the current knowledge on the physiology of balance and on the association between balance deficits and cervical dystonia in other clinical conditions (e.g., whiplash injury), a rationale is therefore offered to a confirmation of the hypothesis that DM1 patients may suffer from cervical ataxia.

The primary endpoint is the demonstration of an association between balance deficits in standing and cervical proprioception deficit in adults affected by Myotonic dystrophy 1.

Secondary endpoints are:

* the investigation of the correlation among the two deficits and the clinical conditions of patients,
* the definition of normative data in the measure of cervical proprioception in a sample of healthy participants.

It is expected that high scores in postural balance, obtained on the posturographic Equitest™-Sensory Organization Test-SOT, correspond to high levels of repositioning accuracy in tests of cervical repositioning and low SOT scores correspond to low accuracy. Moreover, it is expected that an association exists among the two deficits and the clinical situation of the patients. Results from the present pilot study will allow an estimate of the sample size for future experimental protocols. The evidence for an association between balance deficits and cervical ataxia would be of obvious relevance to the patients. This would also support the hypothesis that neck muscle spindles may be especially affected in DM1. This would highlight that muscles are also crucial sensory organs, involved in the perception of joint position, muscle strength, and fatigue. Results from the present study might allow the definition of new rehabilitative programs, such as treatments through a neck strengthening (and thus stiffening) exercise program. This study, therefore, might stimulate new research hypothesis at the neurophysiologic level and possibly lead to findings generalizable from DM1 to other forms of myopathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DM1 since at least 5 years;
* Ability to stand erect with open eyes for at least 20 s;
* Rivermead Mobility Index (RMI) score ≥ 10/15;
* Visual acuity > 10/20, also with corrective lenses;
* Mini Mental State Examination (MMSE) score ≥ 26/30;
* ability to wittingly sign the informed consent form.

Exclusion Criteria:

* neurological or orthopedic pathologies with impact on balance;
* pregnancy;
* previous orthopedic surgical intervention;
* head or neck trauma in the 6 months preceding the study;
* other pathological conditions which could alter balance;
* drug therapy, underway for less than one month before the study, with impact on balance.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The participants will be recruited in the NeuroMuscolar Omniservice (NEMO) clinical centre, on an outpatient basis, from a physiatric referral, or from an inpatient rehabilitation unit.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
SOT score | Day 1
  The patient's task is to maintain an upright stance during 3 20 s trials under six different conditions, including platform and visual surround 'tuned' with individual's sagittal oscillation. The SOT score will be calculated by comparing the sagittal oscillation of the body's centre of mass (COM) to the maximal sagittal oscillation. Score is averaged across the six conditions (range 0 - 100 the higher the score, the lower the oscillation).

SECONDARY OUTCOMES:
Head Repositioning Accuracy, HRA | Day 1
  The head repositioning accuracy in percentage will be computed as the joint position error (JPE) divided by the target position. The JPE will be computed as the absolute difference between the target position and the measured position.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Tesio, MD, Full professor, Principal Investigator — Istituto Auxologico Italiano
Locations (2):
- Italy (2):
  - Istituto Auxologico Italiano, Milan, MI
  - The NEuroMuscular Omnicentre (NEMO) Clinical Center, Milan, MI

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Galli M, Cimolin V, Crugnola V, Priano L, Menegoni F, Trotti C, Milano E, Mauro A. Gait pattern in myotonic dystrophy (Steinert disease): a kinematic, kinetic and EMG evaluation using 3D gait analysis. J Neurol Sci. 2012 Mar 15;314(1-2):83-7. doi: 10.1016/j.jns.2011.10.026. Epub 2011 Nov 25. PMID 22118863
- [Background] Jimenez-Moreno AC, Raaphorst J, Babacic H, Wood L, van Engelen B, Lochmuller H, Schoser B, Wenninger S. Falls and resulting fractures in Myotonic Dystrophy: Results from a multinational retrospective survey. Neuromuscul Disord. 2018 Mar;28(3):229-235. doi: 10.1016/j.nmd.2017.12.010. Epub 2017 Dec 27. PMID 29361394
- [Background] Pieterse AJ, Luttikhold TB, de Laat K, Bloem BR, van Engelen BG, Munneke M. Falls in patients with neuromuscular disorders. J Neurol Sci. 2006 Dec 21;251(1-2):87-90. doi: 10.1016/j.jns.2006.09.008. Epub 2006 Nov 9. PMID 17097113
- [Background] Hammaren E, Kjellby-Wendt G, Kowalski J, Lindberg C. Factors of importance for dynamic balance impairment and frequency of falls in individuals with myotonic dystrophy type 1 - a cross-sectional study - including reference values of Timed Up & Go, 10m walk and step test. Neuromuscul Disord. 2014 Mar;24(3):207-15. doi: 10.1016/j.nmd.2013.12.003. Epub 2013 Dec 15. PMID 24412157
- [Background] Proske U, Gandevia SC. The proprioceptive senses: their roles in signaling body shape, body position and movement, and muscle force. Physiol Rev. 2012 Oct;92(4):1651-97. doi: 10.1152/physrev.00048.2011. PMID 23073629
- [Background] Sansone VA, Lizio A, Greco L, Gragnano G, Zanolini A, Gualandris M, Iatomasi M, Heatwole C. The Myotonic Dystrophy Health Index: Italian validation of a disease-specific outcome measure. Neuromuscul Disord. 2017 Nov;27(11):1047-1053. doi: 10.1016/j.nmd.2017.07.004. Epub 2017 Jul 10. PMID 28890289
- [Background] Tesio L, Alpini D, Cesarani A, Perucca L. Short form of the Dizziness Handicap Inventory: construction and validation through Rasch analysis. Am J Phys Med Rehabil. 1999 May-Jun;78(3):233-41. doi: 10.1097/00002060-199905000-00009. PMID 10340421
- [Background] Tesio L, Rota V, Longo S, Grzeda MT. Measuring standing balance in adults: reliability and minimal real difference of 14 instrumental measures. Int J Rehabil Res. 2013 Dec;36(4):362-74. doi: 10.1097/MRR.0000000000000037. PMID 24185405
- [Background] Beinert K, Taube W. The effect of balance training on cervical sensorimotor function and neck pain. J Mot Behav. 2013;45(3):271-8. doi: 10.1080/00222895.2013.785928. PMID 23663191
- [Background] Loudon JK, Ruhl M, Field E. Ability to reproduce head position after whiplash injury. Spine (Phila Pa 1976). 1997 Apr 15;22(8):865-8. doi: 10.1097/00007632-199704150-00008. PMID 9127919
- [Background] Grip H, Sundelin G, Gerdle B, Karlsson JS. Variations in the axis of motion during head repositioning--a comparison of subjects with whiplash-associated disorders or non-specific neck pain and healthy controls. Clin Biomech (Bristol). 2007 Oct;22(8):865-73. doi: 10.1016/j.clinbiomech.2007.05.008. Epub 2007 Jul 9. PMID 17619066
- [Background] Ferrario VF, Sforza C, Serrao G, Grassi G, Mossi E. Active range of motion of the head and cervical spine: a three-dimensional investigation in healthy young adults. J Orthop Res. 2002 Jan;20(1):122-9. doi: 10.1016/S0736-0266(01)00079-1. PMID 11853078
- [Background] Mortensen JD, Vasavada AN, Merryweather AS. The inclusion of hyoid muscles improve moment generating capacity and dynamic simulations in musculoskeletal models of the head and neck. PLoS One. 2018 Jun 28;13(6):e0199912. doi: 10.1371/journal.pone.0199912. eCollection 2018. PMID 29953539
- [Background] Vasavada AN, Hughes E, Nevins DD, Monda SM, Lin DC. Effect of Subject-Specific Vertebral Position and Head and Neck Size on Calculation of Spine Musculoskeletal Moments. Ann Biomed Eng. 2018 Nov;46(11):1844-1856. doi: 10.1007/s10439-018-2084-9. Epub 2018 Jul 9. PMID 29987540
- [Background] Vasavada AN, Li S, Delp SL. Influence of muscle morphometry and moment arms on the moment-generating capacity of human neck muscles. Spine (Phila Pa 1976). 1998 Feb 15;23(4):412-22. doi: 10.1097/00007632-199802150-00002. PMID 9516695
- [Background] Tesio L. Outcome measurement in behavioural sciences: a view on how to shift attention from means to individuals and why. Int J Rehabil Res. 2012 Mar;35(1):1-12. doi: 10.1097/MRR.0b013e32834fbe89. PMID 22315141